CLINICAL TRIAL: NCT02634944
Title: The Use of the VOMS Tool With Military Personnel to Track Mild Traumatic Brain Injury Recovery and Return to Duty Status
Brief Title: The Use of the VOMS Tool With Military Personnel to Track mTBI Recovery and RTD Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anthony P. Kontos, Ph.D., PhD, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PRO15090054
Record Dates: First submitted 2015-12-03; First posted 2015-12-18 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Concussion; Vestibular; Ocular-Motor
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mTBI (Experimental): mTBI (concussed) participants will be administered the VOMS after concussive event. The VOMS- which requires only a small target with 14 point font text and takes only 5 min to administer- includes assessments in five domains: (1) smooth pursuits, (2) horizontal and vertical saccades, (3) near point of convergence (NPC) distance, (4) horizontal and vertical VOR, and (5) VMS.
  Interventions: Diagnostic Test: Vestibular Ocular Motor Screening Tool (VOMS)
- Healthy Control (Sham Comparator): Healthy controls will be administered the VOMS tool. The VOMS- which requires only a small target with 14 point font text and takes only 5 min to administer- includes assessments in five domains: (1) smooth pursuits, (2) horizontal and vertical saccades, (3) near point of convergence (NPC) distance, (4) horizontal and vertical VOR, and (5) VMS.
  Interventions: Diagnostic Test: Vestibular Ocular Motor Screening Tool (VOMS)
- BLAST mTBI (Experimental): Blast mTBI (concussed) participants will be administered the VOMS after concussive blast event. The VOMS- which requires only a small target with 14 point font text and takes only 5 min to administer- includes assessments in five domains: (1) smooth pursuits, (2) horizontal and vertical saccades, (3) near point of convergence (NPC) distance, (4) horizontal and vertical VOR, and (5) VMS.
  Interventions: Diagnostic Test: Vestibular Ocular Motor Screening Tool (VOMS)
- BLUNT mTBI (Experimental): Blunt mTBI (concussed) participants will be administered the VOMS after concussive blunt event. The VOMS- which requires only a small target with 14 point font text and takes only 5 min to administer- includes assessments in five domains: (1) smooth pursuits, (2) horizontal and vertical saccades, (3) near point of convergence (NPC) distance, (4) horizontal and vertical VOR, and (5) VMS.
  Interventions: Diagnostic Test: Vestibular Ocular Motor Screening Tool (VOMS)

INTERVENTIONS:
Diagnostic Test: Vestibular Ocular Motor Screening Tool (VOMS) — Vestibular Ocular Motor Screening Tool (VOMS)

SUMMARY:
The purpose of the proposed project is to determine if the VOMS is an effective screening tool to identify and track recovery of vestibular and ocular motor impairment and symptoms following mTBI, that corpsman-level medical personnel can successfully implement in combat and non-combat environments. A second purpose of the project is to determine if impairment and symptoms on the VOMS is more pronounced following blast compared to blunt mTBI.

DETAILED DESCRIPTION:
Vestibular impairment and symptoms are prevalent following mild traumatic brain injury (mTBI) and may play a role in prolonged recovery. Researchers have indicated that ocular motor dysfunction and symptoms are common among personnel exposed to blast mTBI. In fact, researchers have suggested that vestibular and ocular motor outcomes such as VOR and vestibulo-spinal reflex (VSR) may be useful in identifying the effects of blast from blunt mTBI. There are currently no brief, clinical screening tools to identify vestibular/ocular motor impairment and symptoms in military personnel following mTBI. Our research team recently developed the Vestibular/Ocular Motor Screening (VOMS) tool to screen for vestibular/ocular motor impairment and symptoms following mTBI. Our preliminary research indicates that VOMS- a 5-min clinical screening tool that can be deployed by corpsman-level (i.e., Special Operation Combat Medics [SOCM], Special Forces Medical Sergeants [18D]) medical personnel with minimal training and materials- was nearly 90% accurate in identifying patients with mTBI from healthy controls. These preliminary findings suggest that VOMS may augment current clinical screening tools- such as the MACE- used by the U.S. Military. The proposed project addresses the "studies to develop standardized metrics for vestibular assessment and monitoring for return to duty" area in the Diagnostics subsection of the Hearing Loss/Dysfunction, Balance Disorder, and or Tinnitus section under the Clinical Trial Research Focus Area.

ELIGIBILITY:
Inclusion Criteria:

* All Participants:

  * Military personnel;
  * Age 18-40 years;
  * Normal or corrected normal vision
* mTBI Participants:

  * Diagnosed with mTBI (blast, blunt, or combo) within past 7 days
  * Clear mechanism of injury
  * Glasgow Coma Scale (GCS) = 13-15
  * Reported or observed signs (Loss of consciousness [LOC], amnesia, disorientation/confusion) at time of injury
  * Current reported symptoms and/or impairment (cognitive, balance, visual)

Exclusion Criteria:

* History of vestibular disorder;
* History of neurological disorder;
* History of previous moderate to severe TBI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 452 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Reliability of US military corpsmen-level medical personnel (i.e., Special Operation Combat Medics [SOCM], Special Forces Medical Sergeants [18D]) to administer the VOMS to US military personnel in combat and non-combat environments. | 6 months
  In-person and telemedicine VOMS (Vestibular Ocular-Motor Screening) training with USASOC medical personnel, followed by repeated VOMS measures to examine reliability of symptom report
Change in symptoms on the VOMS at acute and sub-acute time periods correlated with recovery times to return to duty (RTD) | 3 time periods: 1-7 days post injury; 8 days to 3 months post injury; return to duty (RTD-time period is variable because it is based on individual recovery-assessed up to 36 months)
Reliability of US military corpsmen-level medical personnel (i.e., Special Operation Combat Medics [SOCM], Special Forces Medical Sergeants [18D]) to administer the VOMS to US military personnel in combat and non-combat environments. | 6 months
  In-person and telemedicine VOMS (Vestibular Ocular-Motor Screening) training with USASOC medical personnel, followed by repeated VOMS measures to examine reliability of near point convergence measurements in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Monti, PA, Principal Investigator — First Special Forces Group - JBLM
Locations (1):
- First Special Forces Group - JBLM, Fort Lewis, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited into FITBIR (Federal Interagency Traumatic Brain Injury Research)

REFERENCES:
- [Background] Mucha A, Collins MW, Elbin RJ, Furman JM, Troutman-Enseki C, DeWolf RM, Marchetti G, Kontos AP. A Brief Vestibular/Ocular Motor Screening (VOMS) assessment to evaluate concussions: preliminary findings. Am J Sports Med. 2014 Oct;42(10):2479-86. doi: 10.1177/0363546514543775. Epub 2014 Aug 8. PMID 25106780